CLINICAL TRIAL: NCT07031518
Title: Pilot Study to Identify and Validate Digital Biomarkers in Osteoarthritis of the Knee
Acronym: DigitOAK
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Liege (Other)
Collaborators: Centre Hospitalier Régional de la Citadelle (Other); SYSNAV (Industry)
Responsible Party: Principal Investigator, Margaux POLEUR, Principal Investigator, Neurologist, Centre Hospitalier Universitaire de Liege
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: DigitOAK
Record Dates: First submitted 2025-05-15; First posted 2025-06-22 (Actual); Last update posted 2025-07-30 (Actual); Status verified 2025-07

CONDITIONS: Osteoarthritis of the Knee
Keywords: osteoarthritis of the knee; digital outcome
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patient with osteoarthritis of the knee (Active Comparator): Patients will have two visits: one at inclusion and a second two months later. They will wear Syde® magneto-inertial sensors, one on each ankle, for the month following the initial visit, then a Syde® sensor on the ankle and another on the wrist on the side of the non-dominant hand for the following month. The total duration of the recording period is two months.
  Interventions: Device: Syde; Diagnostic Test: The Self-Paced 40-meter Walk Test (SPWT); Diagnostic Test: 30-second chair stand test (30s-CST); Diagnostic Test: The Timed up and go test (TUG); Diagnostic Test: Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC 3.1); Diagnostic Test: Patient global impression of severity (PGI-S); Other: Pain Level Diary; Other: Qualitative Interview
- Healthy Subjects (Active Comparator): Healthy subjects with similar age and BMI to patients with osteoarthritisof the knee
  Interventions: Device: Syde; Diagnostic Test: The Self-Paced 40-meter Walk Test (SPWT); Diagnostic Test: 30-second chair stand test (30s-CST); Diagnostic Test: The Timed up and go test (TUG)

INTERVENTIONS:
Device: Syde — Actimyo/Syde is an innovative device intended to be used in a home-based environment. It is composed of two watch-like sensors, each containing a magneto-inertial sensors that record the linear acceleration, the angular velocity, the magnetic field of the movement in all directions.The two watches can be worn as wristwatch or placed near the ankle.
Diagnostic Test: The Self-Paced 40-meter Walk Test (SPWT) — Assesses walking speed over a fixed distance by having participants walk as quickly and safely as possible, but without running, along a 40-meter course.
Diagnostic Test: 30-second chair stand test (30s-CST) — It is a simple assessment of lower body strength and endurance. Participants are instructed to stand up and sit down from a chair as many times as possible in 30 seconds.
Diagnostic Test: The Timed up and go test (TUG) — During this standardized test, the subject is observed and timed while he/she rises from a chair, walks 3 meters, performs a 180° turn, walk back toward the chair and sits down.
Diagnostic Test: Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC 3.1) — The WOMAC is a widely used self-administered health status measure for evaluating pain, stiffness, and function in patients with osteoarthritis of the hip or knee. The WOMAC measures three separate dimensions: pain (5 questions), stiffness (2 questions) and function (17 questions).
  Arms: Patient with osteoarthritis of the knee
Diagnostic Test: Patient global impression of severity (PGI-S) — The PGI-S is a patient-reported measure that evaluates the perceived severity of a condition based on a standardized scale, ranging from "none" to "very severe".
  Arms: Patient with osteoarthritis of the knee
Other: Pain Level Diary — Patients will record their specific OAK average pain level during the day using the VAS scale of 0-10 points for one week at the beginning of each month of recording.
  Arms: Patient with osteoarthritis of the knee
Other: Qualitative Interview — This interview is designed to better understand the patient's perspective on the impact of osteoarthritis of the knee on their motor function and to inform the selection of digital tools in upcoming clinical studies.
  Arms: Patient with osteoarthritis of the knee

SUMMARY:
To date, treatment options for knee osteoarthritis remain limited, and their clinical evaluation is complex due to the day-to-day fluctuations in symptoms.

Hospital tests provide a point-in-time measurement that is influenced by various factors (fatigue, recent activity, weather, etc.), making reliable assessment difficult. The aim of the study is to assess the feasibility and acceptability of monitoring actual activity using the Syde® portable device in up to 30 subjects. Numerical variables derived from data collected by Syde® will be compared with conventional on-site clinical assessment criteria and with data from healthy participants, in order to identify a reliable and robust metric, thereby improving treatment evaluation and personalised patient management.

MAIN OBJECTIVES

* Evaluate the use of the device
* Identify numerical variables and determine the optimal time window for evaluation

Patients will have two visits: one at inclusion and a second two months later. They will wear Syde® magneto-inertial sensors, one on each ankle, for the month following the initial visit, then a Syde® sensor on the ankle and another on the wrist on the side of the non-dominant hand for the following month. The total duration of the recording period is two months.

DETAILED DESCRIPTION:
SECONDARY OBJECTIVES

* To assess external validity

  * Spearman correlation coefficient between variables and WOMAC 3.1 scores
  * Spearman correlation coefficient between results and timed tests
  * Spearman correlation coefficient between results and Kellgren-Lawrence grade
* Assess ability to discriminate between groups

  * Difference between patients and healthy participants, and between the 50% of patients with the lowest WOMAC 3.1 score and the 50% with the highest score, and overlap between groups
  * Difference between the three groups of patients according to WOMAC 3.1 score
* Collect qualitative data: Results of qualitative interviews on significant aspects of mobility and device acceptability
* Identify a stiffness index: Ratio between outcome measurements after 0.5 - 1 - 2 or 3 hours of immobility (at least) for 10 minutes and the same outcome measured over the total recording period, excluding the 10-minute intervals.
* Identify the best time of day for recording

  * The metric properties of the different variables will be calculated over the time periods 1-11; 1-10; 1-9; 1-8; 1-7; 1-6; 1-5; 1-4; 1-3; 1-2 and the first hour of the day in order to identify whether morning stiffness accentuates the difference between OAK and healthy participants.
  * The metric properties of the different variables will be calculated over the time periods 2-12; 3-12; 4-12; 5-12; 6-12; 7-12; 8-12; 9-12; 10-12; 11-12 and 12 hours of the day in order to identify whether evening fatigue accentuates the difference between OAK and healthy participants.

ELIGIBILITY:
Inclusion Criteria:

* Patients with bi- or unilateral Knee Osteoarthritis as confirmed by a qualified rheumatologist/orthopaedist or rehabilitation doctor and having had at least one X-ray or MRI for diagnosis confirmation with Kellgren-Lawrence grade minimum 1
* WOMAC 3.1 total score at screening indicating mild, moderate, or severe symptoms in the past 48 hours
* BMI below 35.0 kg/m2

Exclusion Criteria:

* Patients with significant cognitive disorders, limiting the understanding of the exercises to be performed or the presence of apparent communication difficulties hindering the correct collection of data.
* Unable to walk independently (10 meters without any type of external help)
* History of any joint replacement surgery.
* Currently undergoing or had corticosteroid injections within the past 3 weeks.
* Underwent knee surgery in the past 6 months.
* Expecting joint replacement surgery or arthroscopy within 3 months.
* Pregnant women or women planning to become pregnant during the study
* Presence of any other conditions than osteoarthritis (musculoskeletal or neurological) that may affect normal gait. OA in other joints is not considered as an exclusion criterion as long as OAK is the most significant cause of walking impairment.

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-05-14 (Actual); Primary Completion 2025-09-30 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Total Recording Time Over 2 Months | 2 months
  Total number of hours recorded by the Syde® wearable device over a 2-month period.
Median Daily Recording Time | 2 months
  Median number of hours recorded per day by the Syde® device over the 2-month period.
Days to Reach 180 Recording Hours | 2 months
  Number of days required to reach 180 hours of recording, considered the optimal threshold for analysis.
Intra-Class Correlation of Syde® Outcomes | Entire recording period over 2 months
  Intra-Class Correlation (ICC) of each Syde® outcome calculated over slices of x hours (x = 10 to 90) of data per patient to assess reliability.

SECONDARY OUTCOMES:
Correlation Between Syde® Variables and WOMAC 3.1 Scores | Baseline and 2 months
  Spearman correlation between digital variables and WOMAC 3.1 scores at 2 months.
Correlation Between Syde® Variables and Timed Tests | Baseline and 2 months
  Correlation between digital variables and results from 40 m self-paced test, 30 s chair stand test, and timed up and go test.
Correlation Between Syde® Variables and Kellgren-Lawrence Grade | Baseline
  Spearman correlation between digital variables and Kellgren-Lawrence grade.
Discriminative Power of Syde® Variables | Entire recording period over 2 months
  Differences in Syde® outcomes between patients and controls, and among subgroups based on WOMAC 3.1 scores.
Qualitative Interview on Mobility and Usability | Baseline and Month 2
  Qualitative data from interviews exploring mobility limitations, important measures, and impact on daily life.
Stiffness Index Based on Immobility | Entire recording period over 2 months
  Ratio of outcome measures after 0.5-3 hours of immobility (≥10 minutes) compared to full-day values excluding immobility periods.
Optimal Time of Day for Recording | Entire recording period over 2 months
  Metric properties of outcomes calculated for various time windows (e.g., 1-11h, 2-12h) to assess morning stiffness and evening fatigue.

CONTACTS AND LOCATIONS:
Overall Officials: Laurent Servais, MD, PhD, Study Director — Centre Hospitalier Universitaire de Liege
Locations (1):
- Centre de référence des maladies neuromusculaire (CRMN Liège), Hopital de la Citadelle, Liège, Belgium

IPD SHARING:
Plan to Share IPD: Undecided